CLINICAL TRIAL: NCT02137330
Title: Tolerance and Efficacy of the Swallowable Obalon® Gastric Balloons System in Children With Severe Obesity
Brief Title: Obalon in Children With Severe Obesity
Acronym: Obalon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Valerio Nobili, MD, Bambino Gesù Hospital and Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 539/RA; 539/RA Obalon (Registry Identifier: 539/RA, Ethical Commette of Bambino Gesù Children Hospital, Vatican City)
Record Dates: First submitted 2014-05-07; First posted 2014-05-13 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Severe Pediatric Obesity (BMI > 97° pc -According to Centers for Disease Control and Prevention BMI Charts-); Altered Liver Function Tests; Glycemic Intolerance
Keywords: Obalon swallowable intragastric balloons; Severe obesity; Children
MeSH Terms: conditions — Pediatric Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obalon Arm (Experimental): Children swalowed up to 3 intragastric balloons
  Interventions: Device: Swallowable Obalon® Gastric Balloon
- Dietary and lifestyle changes Arm (No Intervention)

INTERVENTIONS:
Device: Swallowable Obalon® Gastric Balloon
  Arms: Obalon Arm

SUMMARY:
The ongoing global rise in the prevalence of overweight and obesity among all ages and among all ethnic groups, figures into a real epidemic phenomenon. This is accompanied by a higher incidence in serious health risks, already present at an early age, "switching-on" the engine towards obesity-related co-morbid diseases and morbid obesity. Weight loss is the only way to avoid systemic and cardiovascular complications of obesity.

Weight loss devices have been recently introduced in bariatric surgery, also in children. They mostly require invasive procedures to be applied. Mini-invasive devices would be needed to obtain weight loss in the pediatric population, since the early age of involved patients.

Obalon intragastric balloons, are swallowable devices. They are filled with liquid or air, and have been used to induce weight loss in obese adults. The investigators aimed to perform a pilot study in pediatrics, and monitor weight loss, metabolic and cardiovascular parameters modifications, after up-to-3 Obalon® Gastric Balloons placement.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 97° pc -CDC BMI charts-

Exclusion Criteria:

* Prevous abdominal surgery
* Functional gastrointestinal motility disorders

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Weight loss (Kg) | 3 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Children Hospital, Rome, Italy, Italy